CLINICAL TRIAL: NCT06851481
Title: A Prospective, Multi-Center, Single-Arm Study to Evaluate the Safety and Performance of the Ladera Medical Suture-Mediated Closure System When Used to Achieve Hemostasis of Common Femoral Arteriotomies in Patients Undergoing Percutaneous Catheter-Based Interventional Procedures (the FASTEN Study)
Brief Title: The Ladera Suture-Mediated Large Bore Closure Study
Acronym: FASTEN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ladera Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLN02002
Record Dates: First submitted 2025-02-24; First posted 2025-02-28 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Vascular Closure; Femoral Arteriotomy Closure

STUDY DESIGN:
Intervention Model Description: Prospective, non-randomized
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- The Ladera LBC System will be used in all participants enrolled in the study (Experimental)
  Interventions: Device: Ladera LBC System

INTERVENTIONS:
Device: Ladera LBC System — Use of the Ladera LBC System to close the femoral arteriotomy

SUMMARY:
This study evaluates the safety and performance of the Ladera Medical suture-mediated large bore closure (LBC) system in gaining post procedure hemostasis in subjects undergoing interventional catheterization procedures using a large-bore procedure sheath.

DETAILED DESCRIPTION:
The Ladera Medical suture mediated large bore closure (LBC) system is a vascular closure device intended for use in catheterization laboratories following percutaneous interventional catheterization procedures that use the retrograde common femoral artery access route for large bore interventional devices. The function of Ladera LBC System is to percutaneously close the puncture in the artery wall (arteriotomy) through which the catheters were inserted for the procedure.

The study is being conducted to demonstrate the safety and performance of the LBC System in achieving hemostasis in femoral arterial access sites in subjects undergoing percutaneous interventional catheterization procedures using a large-bore procedure sheath.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is ≥ 18 years old
2. Patient is scheduled for elective or planned (i.e., not emergent or urgent) percutaneous interventional catheterization procedures involving access through the common femoral artery using 10 to 24 Fr introducer sheaths (i.e., BAV, TAVR/TAVI, PEVAR, TEVAR)
3. Patient is able to undergo emergent vascular surgery if a complication related to the vascular closure necessitates such surgery
4. Patient is willing and able to complete follow-up requirements
5. Patient has the mental capacity to consent for themselves (i.e., does not require the use of a Legally Authorized Representative), and signs a written Informed Consent Form (ICF) prior participating in the study

Exclusion Criteria:

Patients must be EXCLUDED from participation in this study if ANY of the following criteria are met:

Screening / Baseline

1. Prior intra-aortic balloon pump at access site within 30 days of baseline evaluation
2. Patients with severe inflow disease (iliac artery diameter stenosis > 50%) and/or severe peripheral arterial disease (Rutherford Classification 5 or 6), as confirmed with prior standard of care Computed Tomography (CT) Imaging
3. Common femoral artery and iliac lumen diameter is < 6 mm as confirmed with prior standard of care CT Imaging
4. Common femoral artery calcium at the arteriotomy site (i.e., target access site), which is visible with prior CT Imaging
5. Marked tortuosity (at the investigator's discretion) of the femoral or external iliac artery in the target leg based on prior CT Imaging
6. In opinion of the investigator, significant scarring of the target access site which would preclude use of the device in accordance with the IFU
7. Prior target artery closure with any closure device < 90 days, or closure with manual compression ≤ 30 days prior to index procedure
8. Prior atherectomy, vascular surgery, vascular graft, or stent in region of access site
9. Patients receiving glycoprotein IIb/IIIa inhibitors within 24 hours prior to, during, or within 48 hours after the catheterization procedure
10. Patients with significant anemia (Hgb < 9 g/dL, Hct < 30%)
11. Patient with known bleeding disorder including thrombocytopenia (platelet count < 100,000), thrombasthenia, hemophilia or Von Willebrand's disease or known Type II heparin-induced thrombocytopenia
12. Patient with renal insufficiency (serum creatinine level > 221 μmol/L or 2.5 mg/dL), on dialysis therapy, or with renal transplant
13. Known severe allergy to contrast reagent that cannot be managed with premedication
14. Inability to tolerate aspirin and/or other anticoagulation/antiplatelet treatment
15. Planned anticoagulation therapy post-procedure such that ACT is expected to be elevated above 250 seconds for more than 24 hours after the procedure
16. Connective tissue disease (e.g., Marfan's Syndrome)
17. Thrombolytics (e.g., Tissue Plasminogen Activator (t-PA), streptokinase, urokinase), Angiomax (bivalirudin) or other thrombin-specific anticoagulants ≤ 24 hours prior to the index procedure
18. Recent (within 8 weeks) cerebrovascular accident or Q-wave myocardial infarction or acute coronary syndrome (i.e., unstable angina or myocardial infarction) within 48 hours of the index procedure
19. Patients who are morbidly obese (Body Mass Index (BMI) > 40 kg/m2) or cachectic (BMI < 20 kg/m2)
20. Planned major intervention or surgery, including planned interventional catheterization procedure in the target leg, within 30 days following the interventional procedure
21. Patient unable to ambulate at baseline (i.e., confined to wheelchair or bed)
22. Currently participating in a clinical study of an investigational device or drug that has not completed its primary study endpoint
23. Known allergy to any of the materials used in the investigation device (refer to IFU)
24. Patient is known or suspected to be pregnant or lactating or planning to become pregnant within 30 days following the index procedure
25. Evidence of active systemic or local groin infection
26. Patient has other medical, social or psychological problem that in the opinion of the Investigator precludes them from participating
27. Patient is mentally incompetent or a prisoner
28. Patient would refuse blood transfusion if it were to be needed
29. New York Heart Association (NYHA) Class IV heart failure that is uncontrolled and requires treatment in the Intensive Care Unit within 24 hours prior to the index procedure
30. Left Ventricular Ejection Fraction (LVEF) < 20%
31. Unilateral or bilateral lower extremity amputation
32. Known existing nerve damage in the target leg
33. Patients who have already participated in this Investigational study
34. Patients who are currently participating in any other investigational studies Intra-Procedure
35. Patient has a tissue tract (i.e., estimated distance from skin entry point to arterial anterior surface at arteriotomy) expected to be greater than 8 cm
36. Access site above the most inferior border of the IEA and/or above the inguinal ligament based upon bony landmarks
37. Access site in the profunda femoris or superficial femoral arteries, or the bifurcation of these vessels
38. Ipsilateral femoral venous sheath during the catheterization procedure
39. Patient in which there is difficulty inserting the introducer sheath or need for greater than 2 ipsilateral arterial punctures at the start of the catheterization procedure
40. Difficulty in obtaining vascular access resulting in multiple arterial punctures and/or posterior arterial puncture
41. Evidence of a hematoma (> 1.5 cm in diameter), arteriovenous fistula, pseudoaneurysm, or intraluminal thrombosis at the access site
42. Angiographic evidence of arterial laceration, dissection, or stenosis in the femoral artery that would preclude use of the investigational device
43. Index procedural sheath < 10 Fr or > 24 Fr
44. Activated clotting time (ACT) greater than 250 seconds, unless protamine has been administered, immediately prior to index procedure sheath removal and planned vascular closure
45. Uncontrolled hypertension (systolic blood pressure greater than 180 mmHg or diastolic blood pressure greater than 110 mmHg) or hypotension (systolic blood pressure less than 90 mmHg) without pharmacological intervention at the time of index sheath removal and planned vascular closure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2025-08-18 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoint: Major Arterial Access Site Closure-related Complications | 30 days post-procedure
  Freedom from Clinical Events Committee (CEC) adjudicated major complications of the target limb access site within 30 days post-procedure
Primary Performance Endpoint: Time to Hemostasis | Post-procedure, usually within 3 hours
  The mean Time to Hemostasis (TTH) in the Common Femoral Artery (CFA) of the target limb access site with use of the investigational device.

CONTACTS AND LOCATIONS:
Locations (6):
- Australia (3):
  - Jessie McPherson Private Hospital, Clayton, Clayton VIC
  - Macquarie University, Sydney, New South Wales
  - Monash Health, Victoria Heart Hospital, Melbourne, Victoria
- AZ Sint-Jan Brugge AV, Bruges, Belgium
- Netherlands (2):
  - OLVG Amsterdam, Amsterdam
  - Erasmus University Medical Center, Rotterdam

IPD SHARING:
Plan to Share IPD: No